CLINICAL TRIAL: NCT04597268
Title: Safety and Efficacy of Dexmedetomidine vs Ketamine vs Midazolam Combined With Propofol in Gastrointestinal Procedures for Cancer Patients
Brief Title: Dexmedetomidine Versus Ketamine Versus Midazolam in Endoscopic Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Walaa Youssef Elsabeeny, Lecturer of anesthesia and pain management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP2007-50110
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Sedation and Analgesia
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine; Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dexmedetomidine (Experimental): IV dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- ketamine (Experimental): IV ketamine
  Interventions: Drug: Ketamine
- Midazolam (Active Comparator): IV midazolam
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — intravenous dexmedetomidine 1 mic/kg
  Other Names: propofol- dexmedetomidine
  Arms: dexmedetomidine
Drug: Ketamine — ketamine 1mg/kg
  Other Names: propofol- ketamine
  Arms: ketamine
Drug: Midazolam — midazolam 0.05 mg/kg
  Other Names: propofol- midazolam
  Arms: Midazolam

SUMMARY:
This study aims to assess the safety and efficacy of dexmedetomidine versus ketamine versus midazolam combined with propofol in cancer patients undergoing gastrointestinal endoscopic procedures.

DETAILED DESCRIPTION:
Comparison between using intravenous (IV) propofol combined with either IV dexmedetomidine or IV ketamine or IV midazolam; to study the effect of their combination on level of sedation and hemodynamic stability on adult patients scheduled for gastrointestinal endoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for gastrointestinal endoscopic procedures
* ≥ Age 18 years
* ASA I-II

Exclusion Criteria:

* Allergy to any of the used drugs
* impaired renal or liver functions
* hypertensive patients
* patients with cardiovascular
* cerebrovascular disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Ramsy sedation score (RSS) | 3 to 6 months
  time to achievement of Ramsy sedation score (RSS) 3-4, Ramsy sedation scale score from 1 to 6, 1 meaning anxious and 6 meaning no response to stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Y Elsabeeny, MD, Principal Investigator — Lecturer; Nahla Y Shehab, MD, Study Director — Lecturer
Locations (1):
- Walaa Y Elsabeeny, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Data available upon reasonable request through contacting the corresponding author